CLINICAL TRIAL: NCT01637272
Title: A Multi-center, Intra-patient Dose Escalation Phase II Study to Evaluate the Preliminary Efficacy, Safety and Pharmacokinetics of Pasireotide (SOM230) Subcutaneous (s.c.) Followed by Pasireotide LAR in Patients With Dumping Syndrome
Brief Title: Phase II Study Evaluating Efficacy, Safety and Pharmacokinetics of Pasireotide in Patients With Dumping Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230X2203; 2012-001534-34 (EudraCT Number)
Record Dates: First submitted 2012-05-09; First posted 2012-07-11 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Dumping Syndrome
Keywords: Dumping syndrome; SOM230; pasireotide LAR
MeSH Terms: conditions — Dumping Syndrome | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOM230 (Experimental): Subjects with dumping syndrome treated with pasireotide
  Interventions: Drug: SOM230

INTERVENTIONS:
Drug: SOM230 — Pasireotide (SOM230) sc injection was provided as solution for injection in individual 1-point-cut 1 mL ampule, containing nominally 200 μg of pasireotide (as free base). Doses: 50, 100, 150 and 200 μg. Pasireotide im LAR depot injection was provided as micro particles powder in vials containing nominally 10, 20, 40 & 60 mg of pasireotide (as free base) & solvent for suspension for injection in ampules for the reconstitution of the LAR micro particles. Doses: 10, 20, 30, 40 or 60 mg
  Other Names: pasireotide

SUMMARY:
multi-center, phase II study evaluating efficacy, safety and pharmacokinetics of pasireotide in patients with dumping syndrome

DETAILED DESCRIPTION:
43 adult patients with dumping syndrome received pasireotide s.c. during the dose escalation phase (3 months dose could be increased based on the presence of hypoglycemia during OGTT). After completing Month 3, patients were switched to pasireotide LAR for 3 months (up to Month 6). The core phase of the study was completed at the end of Month 6. Patients were allowed to enter the 6 month extension phase if they experienced benefit with pasireotide LAR treatment.

ELIGIBILITY:
Inclusion criteria:.

* Male or female patients ≥ 18 years of age.
* Post-gastric or esophageal bypass surgery, matching one of the criteria below:
* Bariatric surgery: more than 6 months before signing the informed consent
* Esophageal cancer surgery: were disease free at study entry
* Gastric cancer surgery: were at stage 0 or I and were disease free at study entry
* Patient with a documented diagnosis of Dumping Syndrome defined as having:
* History of/or active symptoms associated with dumping syndrome (e.g. post-prandial tachycardia, bloating, diarrhea) and
* Documented history of hypoglycemia based on either:
* glucose <50 mg/dL or 2.8 mmol/L on a sporadic or scheduled blood analysis -or
* glucose value <60 mg/dL or ≤ 3.3 mmol/L at 90, 120, 150 or 180 min during an OGTT
* Patients had at least one glucose level <60 mg/dL (or ≤ 3.3 mmol/L) at 90, 120, 150 or 180 min during the 3-hour OGTT at screening.
* Patients with esophageal cancer with a negative computed tomography (CT) or Magnetic resonance imaging (MRI) scan (neck, thoracic, and upper abdominal) and albumin

  ≥ 3.5 g/dl at baseline.
* Patients with gastric cancer with a negative CT or MRI scan (total abdomen).
* Karnofsky Performance Status ≥ 60 (i.e. required occasional assistance, but was able to care for most of their personal needs)
* Patients who received other therapies for dumping syndrome (such as acarbose, gama guar, pectin) must have stopped all treatments and had a wash out period prior to signing the informed consent (i.e. at least 2 weeks between last previous therapy and first dose of study medication in this study).
* Patients who had provided signed written informed consent prior to study participation.

Exclusion Criteria:

* Bariatric patients who had lap band.
* Patients with a current diagnosis of diabetes mellitus.
* Patients who had failed treatment with somatostatin analogues for dumping syndrome in the past.
* Patients who had been treated with somatostatin analogues in the past, must have had an appropriate interval between the last administration of somatostatin analogues treatment and the study drug as follows
* Octreotide sc for ≥ 72 hours
* Octreotide LAR for ≥ 56 days (8 weeks)
* Lanreotide Autogel for ≥ 98 days (14 weeks)
* Lanreotide SR ≥ 28 days (4 weeks)
* Patients who were already treated with pasireotide.
* Patients who had a known hypersensitivity to somatostatin analogues.
* Patients who were receiving anti-cancer therapy (chemotherapy and/or radiotherapy).
* Patients who had any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunodeficiency, including a positive human immunodeficiency virus (HIV) test result (ELISA and Western blot). An HIV test was not required; however, previous medical history was reviewed.
* Non-malignant medical illnesses that were uncontrolled or whose control may have been jeopardized by the treatment with this study treatment.
* Life-threatening autoimmune and ischemic disorders.
* Patients with the presence of active or suspected acute or chronic uncontrolled infection.

Inadequate end organ function as defined by:

* Inadequate bone marrow function:
* White blood cells (WBC) <2.5 x 109/L
* Absolute neutrophil count <1.5 x 109/L
* Platelets <100 x 109/L
* Hemoglobin <9 g/dL
* International normalized ratio (INR) ≥ 1.3
* Serum creatinine >2.0 mg/dL
* Alkaline phosphatase (ALP) >2.5 x upper limit of normal (ULN)
* Serum total bilirubin >1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2 x ULN
* History of liver disease, such as cirrhosis or chronic active hepatitis B and C.
* Presence of Hepatitis B surface antigen (HbsAg) and/ or presence of Hepatitis C antibody test (anti-Hepatitis C Virus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2015-08-07 (Actual); Study Completion 2015-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- United States (6):
  - Ximed Center for Weight Management Ximed Research, La Jolla, California
  - Stanford University Medical Center SC - SOM230X2203, Stanford, California
  - Mayo Clinic - Rochester Mayo MN, Rochester, Minnesota
  - Montefiore Medical Center CLCZ696B2320, The Bronx, New York
  - Texas Tech University Health Science Center, El Paso, Texas
  - Virginia Endocrinology Research SC, Chesapeake, Virginia
- Belgium (4):
  - Novartis Investigative Site, Bruges, Belgium
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- France (3):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Pierre-Bénite
- Germany (2):
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Würzburg
- Netherlands (2):
  - Novartis Investigative Site, Utrecht, Netherlands
  - Novartis Investigative Site, Groningen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 patients were enrolled as planned; 33 patients completed the core sc phase, 31 patients completed the core LAR phase. Of the 31 patients who completed core LAR phase, 27 patients entered the extension phase. Of the 27 patients who entered the extension phase, 23 patients completed the study.
Pre-assignment Details: All patients underwent an OGTT (75g of glucose) and were evaluated at different time points. If the glucose level was <60 mg/dL at 90, 120, 150 or 180 min during the OGTT and all the other eligibility criteria were met, patients were allowed to start study medication. The study was divided in 2 phases, core phase and extension phase.
Period: Overall Study
Arm/Group | SOM230
Started | 43
Completed sc Phase | 33
Completed Core Phase (sc + LAR) | 31
Entered Extension Phase | 27
Completed Core But Did no Enter Ext.. | 4
Completed | 23
Not Completed | 20
Not completed — Adverse Event | 6
Not completed — Unsatisfactory therapeutic effect | 2
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — completed core, did not enter ext. phase | 4
Not completed — Administrative problems | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: The overall study full analysis set (FAS) consisted of all patients who were enrolled in the study (whether treated or not).
Arm/Group | SOM230
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rate in Plasma Glucose Level
Description: Response rate is defined as percentage of patients with no glucose values < 60 mg/dL at 90,120, 150 and 180 min during the Oral Glucose Tolerance Test (OGTT) at the end of s.c. dose escalation phase
Time Frame: at Month 3 (M3)
Population: The sc full analysis set (sc FAS) consisted of all patients who received at least one dose of pasireotide sc during core sc phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOM230 - 3 Months (sc): Subjects with dumping syndrome treated with pasireotide sc
Arm/Group | SOM230 - 3 Months (sc)
Number analyzed (Participants) | 43
percentage of participants | 60.5 [44.41 to 75.02]

2. Secondary Outcome: Response Rate in Plasma Glucose Level
Description: Response rate is defined as percentage of patients with no glucose values < 60 mg/dL at 90,120, 150 and 180 min during the Oral Glucose Tolerance Test (OGTT) at the end of 6 months (end of LAR/Core phase) and at the end of 12 months (extension phase)
Time Frame: at Month 6 (M6), Month 12 (M12)
Population: The LAR full analysis set (LAR FAS) consisted of all patients who received at least one dose of pasireotide LAR during core LAR phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOM230- 6 Months (LAR): Subjects with dumping syndrome treated with pasireotide sc (3M)followed by pasireotide LAR (3M) for a total of 6 months
- SOM230 - 12 Months (Ext): Subjects with dumping syndrome treated with pasireotide LAR (6 months in Core & 6 months in Ext. phase)
Arm/Group | SOM230- 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 33 | 33
percentage of participants | 36.4 [20.40 to 54.88] | 39.4 [22.91 to 57.86]

3. Secondary Outcome: Response Rate in Pulse Rate
Description: Pulse rate was defined as percentage of patients with change in pulse rate >=10 bpm from pre-OGTT to 30 minutes post OGTT.
Time Frame: at baseline, M3, M6, M12
Population: The sc full analysis set (sc FAS) consisted of all patients who received at least one dose of pasireotide sc during core sc phase. The LAR full analysis set (LAR FAS) consisted of all patients who received at least one dose of pasireotide LAR during core LAR phase.
Measure: Number; unit: Percentage of participants
Groups:
- SOM230 - 6 Months (LAR): Subjects with dumping syndrome treated with pasireotide sc (3M) followed by pasireotide LAR (3M) for a total of 6 months
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 43 | 33 | 33
Percentage of participants
  rate ≥ 10 bpm at baseline | 60.5 | 24.2 | 24.2
  rate ≥ 10 bpm at post-baseline | 18.6 | 36.4 | 27.3

4. Secondary Outcome: Response Rate in Hematocrit Levels
Description: Percentage of patients with change in hematocrit >= 3% from pre-OGTT to 30 minutes post OGTT.
Time Frame: M3, M6, M12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 43 | 33 | 33
Percentage of participants
  hematocrit >= 3% at baseline | 27.9 | 21.2 | 21.2
  hematocrit >= 3% at post baseline | 16.3 | 27.3 | 24.2

5. Secondary Outcome: Insulin Levels During OGTT
Description: Absolute insulin levels at the end of M3, M6, M12
Time Frame: M3, M6, M12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 43 | 33 | 33
pmol/L
  Pre-OGTT (n= 31, 29, 21) | 37.0 (24.55) | 34.7 (19.73) | 29.0 (14.43)
  30 Minutes (n=30, 29, 23) | 196.3 (253.10) | 499.8 (276.80) | 294.1 (177.25)
  60 Minutes (n= 31, 30, 22) | 367.5 (354.73) | 573.2 (428.46) | 602.1 (381.6)
  90 Minutes (n=31, 30, 22) | 309.1 (263.92) | 420.4 (544.78) | 472.0 (438.82)
  120 Minutes(n=32, 30, 22) | 183.7 (209.90) | 205.7 (514.45) | 195.1 (247.43)
  150 Minutes(n=33, 30, 22) | 103.2 (166.67) | 102.8 (228.92) | 76.0 (106.05)
  180 Minutes (n=32, 29, 22) | 58.5 (52.65) | 69.1 (154.11) | 52.0 (58.81)

6. Secondary Outcome: Glucagon Levels During OGTT
Description: Absolute glucagon levels at the end of Months 3, 6 & 12
Time Frame: M3, M6, M12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 43 | 33 | 33
pmol/L
  Pre-OGTT (n= 31, 30, 23) | 20.70 (6.162) | 22.6 (5.85) | 21.4 (6.82)
  30 Minutes (n= 33, 29, 22) | 20.64 (7.037) | 25.8 (6.57) | 23.8 (6.97)
  60 Minutes (n= 33, 28, 22) | 20.80 (7.330) | 23.7 (5.76) | 22.9 (7.07)
  90 Minutes (n= 32, 29, 22) | 20.07 (7.898) | 22.7 (5.16) | 21.5 (7.69)
  120 Minutes (n= 32, 29, 22) | 19.73 (7.369) | 23.1 (5.40) | 22.0 (7.31)
  150 Minutes (n= 32 28, 22) | 19.94 (7.169) | 23.7 (6.67) | 21.8 (7.27)
  180 Minutes (n= 32, 29, 22) | 20.16 (7.097) | 22.7 (5.45) | 22.3 (6.58)

7. Secondary Outcome: Glucagon-like Peptide 1 (GLP-1) Levels During OGTT
Description: Absolute Glucagon-like peptide 1 (GLP-1) levels at the end of at the end of Months 3, 6 and 12 at different time points.
Time Frame: M3, M6, M12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 43 | 33 | 33
pmol/L
  Pre-OGTT (n=31, 29, 23) | 3.021 (2.1936) | 2.1 (1.37) | 1.6 (1.26)
  30 Minutes(n=32, 29, 22) | 12.811 (6.6194) | 21.0 (18.01) | 17.4 (17.64)
  60 Minutes (n= 32, 30, 22) | 11.208 (11.1218) | 14.6 (18.44) | 12.6 (8.76)
  90 Minutes (n=31, 29, 22) | 6.986 (4.9729) | 8.2 (4.96) | 7.2 (3.71)
  120 Minutes (n=31, 29, 22) | 5.003 (4.1183) | 5.2 (3.94) | 5.0 (2.98)
  150 Minutes(n=31, 29, 22) | 3.565 (2.3879) | 4.2 (4.20) | 3.7 (2.46)
  180 Minutes (n=31, 29, 22) | 2.974 (1.9902) | 3.3 (3.49) | 3.2 (2.44)

8. Secondary Outcome: Gastric Inhibitory Polypeptide (GIP) Levels at During OGTT
Description: Absolute Gastric Inhibitory Polypeptide (GIP) levels at the end of Months 3, 6 and 12 at different time points.
Time Frame: M3, M6, M12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 43 | 33 | 33
pmol/L
  Pre-OGTT (n=31, 29, 23) | 2.608 (1.7441) | 1.5 (1.00) | 1.7 (1.51)
  30 Minutes (n=32, 29, 22) | 15.704 (10.6395) | 30.3 (19.73) | 24.8 (18.88)
  60 Minutes (n= 32, 30, 22) | 9.471 (6.1861) | 14.3 (13.37) | 11.6 (9.05)
  90 Minutes(n=31, 29, 22) | 4.141 (2.8978) | 6.5 (7.32) | 5.2 (5.18)
  120 Minutes (n=31, 29, 22) | 2.089 (1.4681) | 2.4 (1.73) | 3.0 (2.81)
  150 Minutes (n=30, 29, 22) | 1.376 (1.2049) | 2.1 (3.22) | 1.9 (1.44)
  180 Minutes (n=31, 29, 22) | 1.260 (1.2218) | 3.8 (12.77) | 2.5 (3.72)

9. Secondary Outcome: Health-related Quality of Live (HRQoL) Short Form- 36 (SF-36) Score(s)
Description: Absolute HRQoL SF-36 Scores at end of the Months 3, 6 and 12 from s.c. baseline. SF-36, a 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting. Items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: M3, M6, M12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 43 | 33 | 33
scores on a scale
  Physical Component Summary (n=35, 29, 23) | 44.801 (8.3378) | 45.306 (9.5622) | 46.505 (8.5105)
  Mental Component Summary (n=35, 29, 23) | 44.093 (12.2144) | 44.838 (11.6573) | 47.021 (11.5053)

10. Secondary Outcome: Dumping Severity Score (DSS) at the End of Months 3, 6 and 8
Description: Absolute Dumping Severity Score (DSS) scores at end of M3, M6 & M8. At study start patients were assessed using DSS (older version of DSQ); however after the implementation of protocol amendment 2, all patients were expected to use DSQ. No results available for M12 as last patient that answered the DSS was at M8. DSS = disease-specific patient (Pt.) reported outcome (PRO) questionnaire uses a 4-point Likert scale (0, absent; 1, mild; 2, relevant; 3, severe; 4) to ask Pt. to evaluate intensity of early dumping symptoms (within 30 minutes (<30 minutes) after food ingestion). The questionnaire also evaluates 65 late dumping symptoms (more than 1.5 hours (>90 minutes) after food ingestion). Early & late dumping score calculated by adding the scores of the respective questions. Cumulative dumping score is obtained by adding early & late scores. DSS Range (min (absent) - max (severe)): Early dumping: 0-24; Late Dumping: 0-18; Cumulative: 0-42. Lower scores represent a better outcome.
Time Frame: M3, M6, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- SOM230 - 8 Months (Ext): Subjects with dumping syndrome treated with pasireotide LAR (6 months in Core & 6 months in Ext. phase)
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 8 Months (Ext)
Number analyzed (Participants) | 43 | 33 | 33
scores on a scale
  Early symptoms (n=20, 9, 2) | 7.1 (6.38) | 6.8 (6.46) | 9.0 (8.49)
  Late symptoms (n=20, 9, 2) | 6.7 (5.42) | 6.4 (5.27) | 6.0 (4.24)
  Overall score (n=20, 9, 2) | 13.7 (11.11) | 13.2 (10.65) | 15.0 (12.73)

11. Secondary Outcome: Dumping Score Questionnaire (DSQ) at the End of Months 3, 6 and 12
Description: Absolute Dumping Score Questionnaire (DSQ) scores at end of Months 3, 6 & 12 from s.c. baseline. DSQ = disease-specific PRO scale. The questionnaire uses a 5-point Likert scale (0, none; 1, mild; 2, moderate; 3, severe; 4, very severe) to ask Pt. to evaluate intensity of 10 early dumping symptoms (within 30 minutes (<30 minutes) after food ingestion). The questionnaire also evaluates 5 late dumping symptoms (more than 1.5 hours (>90 minutes) after food ingestion). Early & late dumping score calculated by adding the scores of respective questions. A cumulative dumping score is obtained by adding early & late scores. At study start patients were assessed using DSS (older version of DSQ); however after the implementation of protocol amendment 2, all patients used DSQ. DSQ Range: (min (None) - max (Very severe)): Early dumping: 0-40; Late Dumping: 0-20; Cumulative: 0-60. Lower scores represent a better outcome.
Time Frame: M3, M6, M12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 43 | 33 | 33
scores on a scale
  Early symptoms (n=15, 20, 23) | 9.6 (10.27) | 9.2 (10.05) | 10.7 (10.94)
  Late symptoms (n=15, 20, 23) | 4.9 (5.37) | 5.6 (6.57) | 5.7 (5.93)
  Overall score (n=15, 20, 23) | 14.5 (15.26) | 14.8 (14.65) | 16.3 (16.23)

12. Secondary Outcome: Patient Global Assessment at the End of Months 3, 6 and 12
Description: Treatment with pasireotide LAR (both early and late dumping scores), was assessed by patient global assessment. Patient Global Assessment served as an additional approach to symptom based measurement by DSQ. It incorporated a patient global assessment question: "Considering all the ways that your disease affects you, rate how you are feeling during the last 7 days compared with your situation before starting the study" .Patients Global Assessment was measured utilizing a 7 point scale (from 1=a lot worse to 7= a lot better).
Time Frame: M3, M6, M12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | SOM230 - 3 Months (sc) | SOM230 - 6 Months (LAR) | SOM230 - 12 Months (Ext)
Number analyzed (Participants) | 35 | 29 | 23
scores on a scale | 5.1 (1.19) | 5.1 (1.27) | 5.9 (0.95)

13. Secondary Outcome: Plasma Pharmacokinetic (PK) Parameter of Pasireotide: Cmax, ss (Steady State) and Ctrough, ss, After s.c. Injection
Description: A pre-dose PK blood sample was collected before the morning pasireotide s.c. dose of 50 μg, 100 ug, 150 ug and 200 ug. OGTT was performed right after the morning s.c. dose (Time point zero); additional PK blood samples were collected at the same time points as the OGTT evaluation at 30, 60, 90, 120, 150 and 180 minutes. 'n' = number of subjects with non-missing values
Time Frame: M1 to M3
Population: The sc PK analysis set consisted of all patients who received at least one of the scheduled full daily sc dose (3 injections) and had evaluable PK data (concentration) in the sc dose escalation phase of the study (Visit 2 through Visit 8).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- SOM sc 50 ug t.i.d.: Subjects with dumping syndrome treated with pasireotide sc 50 ug t.i.d. for 3 months
- SOM sc 100 ug t.i.d.: Subjects with dumping syndrome treated with pasireotide sc 100 ug t.i.d. for 3 months
- SOM sc 150 ug t.i.d.: Subjects with dumping syndrome treated with pasireotide sc 150 ug t.i.d. for 3 months
- SOM sc 200 ug t.i.d.: Subjects with dumping syndrome treated with pasireotide sc 200 ug t.i.d.
Arm/Group | SOM sc 50 ug t.i.d. | SOM sc 100 ug t.i.d. | SOM sc 150 ug t.i.d. | SOM sc 200 ug t.i.d.
Number analyzed (Participants) | 40 | 31 | 23 | 14
ng/mL
  Cmax, ss (n=35, 28, 18, 10) | 1.49 (0.613) | 3.31 (1.78) | 4.56 (2.22) | 5.62 (3.18)
  Ctrough, ss (n=37, 30, 22, 12) | 0.574 (0.436) | 1.11 (0.909) | 1.5 (0.798) | 2.03 (1.54)

14. Secondary Outcome: Plasma Pharmacokinetic (PK) Parameter of Pasireotide: AUC0-3h, ss, After s.c. Injection
Description: A pre-dose PK blood sample was collected before the morning pasireotide s.c. dose of 50 μg, 100 ug, 150 ug and 200 ug. OGTT was performed right after the morning s.c. dose (Time point zero); additional PK blood samples were collected at the same time points as the OGTT evaluation at 30, 60, 90, 120, 150 and 180 minutes.
Time Frame: M1 to M3
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | SOM sc 50 ug t.i.d. | SOM sc 100 ug t.i.d. | SOM sc 150 ug t.i.d. | SOM sc 200 ug t.i.d.
Number analyzed (Participants) | 36 | 28 | 18 | 10
hr*ng/mL | 3.04 (1.13) | 6.53 (3.45) | 8.84 (3.89) | 11.5 (6.23)

15. Secondary Outcome: Plasma Pharmacokinetic (PK) Parameter of Pasireotide: Tmax, ss, After s.c. Injection
Description: as for outcome 14
Time Frame: M1 to M3
Population: as for outcome 13
Measure: Median (Full Range); unit: hr
Arm/Group | SOM sc 50 ug t.i.d. | SOM sc 100 ug t.i.d. | SOM sc 150 ug t.i.d. | SOM sc 200 ug t.i.d.
Number analyzed (Participants) | 36 | 28 | 20 | 11
hr | 0.583 (NA) [0 to 1.58] | 0.6 (NA) [0 to 2.1] | 0.583 (NA) [0.5 to 2.6] | 0.633 (NA) [0.5 to 1.22]

16. Secondary Outcome: Plasma PK Parameter of AUC0-3h, d21, End _inj and AUC0-3h, d28, 3rd_inj Associated With LAR (LAR Core Phase)
Time Frame: M4 to M6
Population: The LAR PK analysis set consisted of all patients who received at least one of the scheduled full monthly im LAR injections and had evaluable PK data (concentration) in the LAR phase of the study (Visit 9 through end of LAR phase visit).
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- SOM LAR 10mg: Subjects with dumping syndrome treated with pasireotide LAR 10mg
- SOM LAR 20mg: Subjects with dumping syndrome treated with pasireotide LAR 20mg
Arm/Group | SOM LAR 10mg | SOM LAR 20mg
Number analyzed (Participants) | 14 | 19
hr*ng/mL
  AUC0-3h,d21, 2nd injection (n = 12, 14) | 6.92 (4.12) | 14.9 (6.71)
  AUC0-3h,d28, 3rd_injection (n = 9, 16) | 5.97 (2.41) | 9.3 (4.11)

17. Secondary Outcome: Summary of LAR PK Parameters by Dose
Description: Summary of plasma PK parameter Cmax, p2 , 2nd injection and Ctrough, d28 associated with LAR injection (LAR Core phase)
Time Frame: M4 to M6
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOM LAR 10mg | SOM LAR 20mg
Number analyzed (Participants) | 14 | 19
ng/mL
  Cmax, p2, 2nd_inj (n = 10, 13) | 3.2 (1.55) | 6.2 (2.6)
  Ctrough (n= 14, 19) | 2.29 (1.05) | 3.33 (1.34)

18. Secondary Outcome: Pasireotide Concentrations in LAR Phase
Description: Summary of pasireotide concentrations following monthly i.m. injections of pasireotide LAR by incident dose (LAR Pharmacokinetic set)
Time Frame: M7 to M12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- SOM LAR 30mg: Subjects with dumping syndrome treated with pasireotide LAR 30mg
- SOM LAR 40mg: Subjects with dumping syndrome treated with pasireotide LAR 40mg
- SOM LAR 60mg: Subjects with dumping syndrome treated with pasireotide LAR 60mg
Arm/Group | SOM LAR 10mg | SOM LAR 20mg | SOM LAR 30mg | SOM LAR 40mg | SOM LAR 60mg
Number analyzed (Participants) | 6 | 12 | 17 | 9 | 3
ng/mL
  M7 - 0hr (pre-dose) (n = 4, 11, 11, 0, 0) | 2.25 (1.56) | 4.3 (2.19) | 7.76 (4.31) | NA (NA) — N/A = No participants took this dose hence no data | NA (NA) — N/A =No participants took this dose hence no data
  M8 - 0hr (pre-dose) (n = 5, 7, 11, 0, 0) | 2.91 (2.42) | 3.77 (1.57) | 6.5 (2.91) | NA (NA) — N/A = No participants took this dose hence no data | NA (NA) — N/A = No participants took this dose hence no data
  M9 - 0hr (pre-dose) (n = 5, 6, 9, 6, 0) | 2.97 (1.68) | 4.01 (2.27) | 6.38 (3.15) | 7.53 (4.45) | NA (NA) — N/A = No participants took this dose hence no data
  M10 - 0hr (pre-dose) (n = 5, 6, 8, 5, 0) | 3.53 (1.75) | 5.48 (3.62) | 8.38 (2.81) | 11.8 (8.26) | NA (NA) — N/A = No participants took this dose hence no data
  M11 - 0hr (pre-dose) (n = 5, 4, 8, 4, 3) | 3.45 (1.98) | 3.48 (0.772) | 7.99 (3.54) | 6.53 (1.83) | 17.9 (7.15)
  M12 - 0hr (pre-dose) (n = 5, 3, 8, 4, 3) | 3.27 (2.02) | 4.63 (1.04) | 10.3 (6.05) | 6.55 (2.05) | 18.1 (13.8)

19. Secondary Outcome: LAR PK Parameter: Ctrough - at Steady State (ss) by Dose
Description: In the LAR treatment phase, monthly injections of pasireotide LAR 10, 20, 30 and 40 mg were given to participants and trough concentration at steady state (Ctrough,ss) were obtained but due to only 1 participant in the 40mg arm, standard deviation could not be calculated.
Time Frame: M4 to M12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOM LAR 10mg | SOM LAR 20mg | SOM LAR 30mg | SOM LAR 40mg
Number analyzed (Participants) | 6 | 6 | 6 | 1
ng/mL | 3.34 (1.52) | 3.76 (1.48) | 8.19 (3.22) | 4.63 (NA) — N/A - due to only one participant at LAR 40 mg, Ctrough,ss for this arm was not enough to a standard deviation

ADVERSE EVENTS:
Groups:
- s.c. Phase: s.c. phase was made up of subjects with dumping syndrome who entered the study and were treated with pasireotide s.c.
- LAR Phase: LAR phase was made up of subjects with dumping syndrome who completed the s.c. phase, entered the LAR phase and were treated with pasireotide LAR
Arm/Group | s.c. Phase | LAR Phase
Serious Adverse Events (participants affected / at risk) | 6/43 | 10/33
Other Adverse Events (participants affected / at risk) | 31/43 | 25/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | s.c. Phase (N=43) | LAR Phase (N=33)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | s.c. Phase (N=43) | LAR Phase (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 3 | 0
Palpitations (Cardiac disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 6 | 6
Steatorrhoea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 5 | 4
Chills (General disorders) | 1 | 2
Fatigue (General disorders) | 3 | 8
Injection site pain (General disorders) | 4 | 1
Injection site reaction (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 0 | 2
Thirst (General disorders) | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 5
Bronchitis (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 6
Sinusitis (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Weight increased (Investigations) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4
Dizziness (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 10 | 9
Syncope (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2
Haematoma (Vascular disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
All safety parameters were analyzed by study phase (sc/LAR)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.